CLINICAL TRIAL: NCT03447665
Title: Infant Behavioral Sleep Intervention: Comparative Efficacy Across Two Approaches "The Sleeping Baby Study"
Brief Title: Infant Behavioral Sleep Intervention: Comparative Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Purdue University (Other); Saint-Joseph University (Other)
Responsible Party: Principal Investigator, Sarah Honaker, Assistant Professor of Pediatrics, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VFR-43-Honaker
Record Dates: First submitted 2018-02-09; First posted 2018-02-27 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Insomnia
Keywords: Infant behavioral sleep intervention; Infant sleep; Pediatric insomnia; Infant night wakings
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Families are randomly assigned to one of three groups: control, bedtime only (intervention), or all night (intervention).
Who Masked: Outcomes Assessor
Masking Description: The individuals coding videosomnography are blinded to the participant's condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Infant sleep monitoring and parental surveys only
- Intervention (Bedtime only) (Experimental): Infant behavioral sleep intervention implemented at bedtime only. Parents are instructed to soothe/help their infant back to sleep after night wakings. Includes a tailored sleep schedule and bedtime routine, as well as support from a sleep interventionist.
  Interventions: Behavioral: Bedtime routine; Behavioral: Sleep schedule; Behavioral: Intervention (bedtime)
- Intervention (All night) (Experimental): Infant behavioral sleep intervention implemented at bedtime and after each subsequent infant night waking. Includes a tailored sleep schedule and bedtime routine, as well as support from a sleep interventionist.
  Interventions: Behavioral: Bedtime routine; Behavioral: Sleep schedule; Behavioral: Intervention (bedtime); Behavioral: Intervention (after night wakings)

INTERVENTIONS:
Behavioral: Bedtime routine — Tailored bedtime routine
  Arms: Intervention (All night); Intervention (Bedtime only)
Behavioral: Sleep schedule — Tailored sleep schedule, including morning rise time, cut-off for last nap of the day, and bedtime.
  Arms: Intervention (All night); Intervention (Bedtime only)
Behavioral: Intervention (bedtime) — Parents implement behavioral sleep intervention at bedtime.
  Arms: Intervention (All night); Intervention (Bedtime only)
Behavioral: Intervention (after night wakings) — Parents implement behavioral sleep intervention following each night waking.
  Arms: Intervention (All night)

SUMMARY:
While frequent night awakenings in newborns are common and expected, an estimated 20-30% of older infants and toddlers have frequent problematic night wakings requiring parental intervention throughout the night. Standard infant behavioral sleep intervention approaches, which require parental intervention throughout the night, are effective but often difficult for families to implement. The aim of this study is to compare the efficacy of two infant behavioral sleep interventions with a no treatment condition, on infant sleep and family functioning. Healthy infants between the ages of 6 and 18 months with night wakings will be randomized into one of three conditions: Entire night intervention, bedtime only intervention, or no treatment.

DETAILED DESCRIPTION:
Study Design: Randomized controlled trial (RCT). Approximately thirty participants will be randomized to a control condition or one of two intervention conditions.

Participants: Participants are healthy infants between the ages of 6 and 18 months who wake during the night, and their parents. Parents must be willing to engage in infant behavioral sleep intervention.

Study Procedure: Participant recruitment strategies include direct referrals from community primary care providers (PCP)s, signs posted in medical offices, and social media posts. Participants will be screened and consented via phone. Team members will conduct three home visits with participating families to install videorecording device and actigraphy and take a sleep history (Visit 1); teach families the intervention (Visit 2); and remove monitoring equipment and offer intervention to families in the control condition (Visit 3). Parents will be asked to complete daily sleep logs and three sets of surveys using REDCap.

Intervention: The intervention consists of an infant behavioral sleep protocol. For both intervention conditions an interventionist will collaborate with the family to design a tailored sleep schedule and bedtime routine. The interventionist will then teach the family a behavioral approach, which involves placing the infant in his/her crib awake, and leaving the room. The behavioral approach will be individually tailored for each family (e.g., periodic checks). The two intervention conditions differ in regards to the timing of the intervention. In the all night condition, which represents a standard intervention approach, parents are asked to implement the behavioral protocol at bedtime and at subsequent night wakings. In the bedtime only condition, parents are asked to implement the behavioral protocol at bedtime only, and to soothe their infant back to sleep following night wakings.

Measures: Infant sleep will be assessed via parent-report (sleep diary and validated measure); actigraphy; and videosomnography. Parent sleep, parent mood, and infant mood will be assessed via validated parental-report survey measures.

Collaborators on this study include: AJ Schwichtenberg, Purdue University; Jodi Mindell, Saint Joseph University.

ELIGIBILITY:
Inclusion Criteria:

* Infant has disruptive night wakings (wakes 1x or more/night, 5+ nights per wk; caregiver intervenes at night wakings)
* Infant is placed in bed asleep in a crib/bassinet or similar at bedtime at least five nights per week
* Parent/caregiver goal is for the infant to fall asleep independently at bedtime and/or return to sleep independently during the night
* Parent/caregiver goal is for the infant to sleep in crib or similar
* Parent/caregiver lives in the home with the infant, is typically at home at the time of the infant's typical bedtime at least 5 nights a week, and is primary caregiver at bedtime and during the night.
* The family must have in-home private wireless access that they are willing to share with the study team (necessary for streaming video)
* Families lives in Indianapolis, Indiana or surrounding areas (within 50 miles of Indiana University School of Medicine)

Exclusion Criteria:

* Infant has a chronic major medical condition that affects sleep
* Infant has a major developmental condition (e.g. Down syndrome)
* Family is already receiving professional help for the infant's sleep problems
* Infant snores 5+ nights per week (in which case a sleep study will be recommended; families could participate in the study following a negative sleep study.)
* Infant has chronic skin conditions (e.g. eczema) that would prohibit wearing an actigraph on the leg

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
Infant sleep (subjective) | Change in score from baseline (day 2, prior to the start of intervention) to post-intervention (day 16)
  Total score on Infant Sleep Questionnaire (ISQ; range=0-38; higher score indicate more problematic sleep)

SECONDARY OUTCOMES:
Infant sleep (objective): wake after sleep onset | Average per night from nights 1-3 (baseline) compared to average from nights 15-17 (2 weeks later; after intervention)
  Wake after sleep onset in minutes (assessed via videosomnography)
Infant sleep (subjective): wake after sleep onset | Average per night from nights 1-3 (baseline) compared to average from nights 15-17 (2 weeks later; after intervention)
  Wake after sleep onset in minutes (assessed via parent report on sleep diary)
Infant sleep (objective): longest sleep period | Average per night from nights 1-3 (baseline) compared to average from nights 15-17 (2 weeks later; after intervention)
  Longest sleep period in minutes (assessed via videosomnography)
Infant sleep (subjective): longest sleep period | Average per night from nights 1-3 (baseline) compared to average from nights 15-17 (2 weeks later; after intervention)
  Longest sleep period in minutes (assessed via parent report on sleep diary)
Parental stress | Average from nights 1-3 (baseline) compared to average from nights 15-17 (2 weeks later; after intervention)
  Daily parental rating of nightly stress associated with their infant's sleep
Parental mood | Baseline (day 2, prior to the start of intervention) compared to post-intervention (day 16)
  Profile of Mood State - 2nd edition, total score
Parental sleep | Baseline (day 2, prior to the start of intervention) compared to post-intervention (day 16)
  Pittsburgh Sleep Quality Index, total score

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided